CLINICAL TRIAL: NCT06653842
Title: A Phase 2, Baseline-Controlled Study Evaluating the Safety and Efficacy of PTX-022 (Sirolimus) Topical Gel 3.9% in the Treatment of Cutaneous Venous Malformations
Acronym: TOIVA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALV-10
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Venous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-arm, open-label (Experimental)
  Interventions: Drug: QTORIN 3.9% rapamycin anhydrous gel

INTERVENTIONS:
Drug: QTORIN 3.9% rapamycin anhydrous gel — QTORIN 3.9% Rapamycin Anhydrous Gel

SUMMARY:
A Phase 2, Baseline-Controlled Study Evaluating the Safety and Efficacy of PTX022 (sirolimus) Topical Gel 3.9% in the Treatment of Cutaneous Venous Malformations

ELIGIBILITY:
Inclusion Criteria: The participant must have a clinically confirmed superficial/ cutaneous (visible on the skin) venous malformation (cVM), referred to as the treatment area. The treatment area may contain a minority (<30%) lymphatic component (mixed venous / lymphatic malformation).

-

Exclusion Criteria:

* The participant's treatment area is mainly in any wet mucosa or within the orbital rim. For clarification, no part of the venous malformation should be evaluated or treated if it in mucosa. External genital presentation is permitted.
* The participant has a known pervasive extension of the lesion into mucosa, bone or tissue (as determined by diagnostic or the investigator) that would impair the ability of the investigator to evaluate the cutaneous components of the lesion.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Week 12

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (cVM-IGA) From Baseline to Week 12 | Change from baseline to Week 12
  Likert scale used by clinicians to evaluate the overall change of the study designated venous malformation
Overall Patient Global Impression of Change (PGI-C) From Baseline to Week 12 | Change from baseline to Week 12
  Likert scale used by patients to evaluate the overall change of the study designated venous malformation

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Children's Hospital of Orange County, Irvine, California
  - Stanford University, Palo Alto, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Johns Hopkins, Baltimore, Maryland
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — https://www.toivatrial.com/